CLINICAL TRIAL: NCT00550498
Title: Phase 1 Study of Bone Marrow - Derived Stem Cell in the Treatment of Ocular Lesions of Behcet's Disease
Brief Title: Stem Cell Transplantation in Ocular Lesions of Behcet's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No improvement obtained in 3 cases. Retinal detachment observed in 2 cases
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3086
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Retinitis; Behcet's Syndrome
Keywords: Retinal Vasculitis; Retinal Edema; Behcet's Disease
MeSH Terms: conditions — Retinitis; Behcet Syndrome; Retinal Vasculitis; Papilledema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Behcet's Disease with ocular lesions
  Interventions: Biological: Autologous Stem Cell Transplantation

INTERVENTIONS:
Biological: Autologous Stem Cell Transplantation — Autologous bone marrow aspiration (20 ml) from iliac crest. Separation of mononuclear cells using ficoll hypaque and culture in 10% fetal bovine serum and Dulbecco modified eagles medium. After confluent stage, detachment of cells with trypsin/EDTA, and subculture. Repeated passages until obtainment of required cell number. Confluent cells of last passage are washed with tyrode solution and incubate with M199 for 60 minutes. Cells are separated using trypsin/EDTA and washed 3 times with M199 and 1% HSA. Precipitate will be diluted with heparinized M199 to make solution with 6×106 cells /ml. Sample will be tested for viability and detection of CD45, CD34, CD90, CD44, CD13, CD105, and CD166 before injection. The number of cells for injection will be between 3-5 million cells, in a maximum volume of 0.3 ml. Cells will be injected in vitreal at 3.5 millimeter of limbus with a 26 gauge insulin needle.

SUMMARY:
The purpose of this study is to find if autologous stem cell transplantation can stop the progression of intractable eye lesions of Behcet's Disease or even to improve it.

DETAILED DESCRIPTION:
To test in a pilot study the effect of autologous stem cell transplantation in stopping the progression of retinal damage of eye lesions in Behcet's Disease by repairing the vascular damage, and possibly to improve the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Behcet's Disease
* Fulfilling the International Criteria for behcet's Disease (ICBD)
* Ocular lesions with retinal vasculitis
* Resistant to at least 3 months of combination therapy with pulse cyclophosphamide (1g/monthly), azathioprine (3 mg/kg/daily), and prednisolone 0.5 mg/kg/daily
* Visual acuity not less than 4 meters finger count
* Retinal edema confirmed by color photography and OCT

Exclusion Criteria:

* No Vision
* Active posterior uveitis
* Fundus not visible

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
1- Visual acuity by ETDRS (Early Treatment of Diabetic Retinopathy Study). 2- Retinal state and retinal edema by Color Photography, Multifocal Electroretinography, and OCT (Optic Coherent Tomography). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, MD, Study Chair — Rheumatology Research Center, Medical Sciences/University of Teheran; Hormoz Shams, MD, Principal Investigator — Rheumatology Research Center, Medical Sciences/University of Tehran; Behrouz Nikbin, MD, Principal Investigator — Department of Immunology, Medical Sciences/University of Tehran
Locations (1):
- Rheumatology Research Center, Behcet's Disease Unit (Shariati Hospital), Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Otani A, Dorrell MI, Kinder K, Moreno SK, Nusinowitz S, Banin E, Heckenlively J, Friedlander M. Rescue of retinal degeneration by intravitreally injected adult bone marrow-derived lineage-negative hematopoietic stem cells. J Clin Invest. 2004 Sep;114(6):765-74. doi: 10.1172/JCI21686. PMID 15372100
- [Background] Kicic A, Shen WY, Wilson AS, Constable IJ, Robertson T, Rakoczy PE. Differentiation of marrow stromal cells into photoreceptors in the rat eye. J Neurosci. 2003 Aug 27;23(21):7742-9. doi: 10.1523/JNEUROSCI.23-21-07742.2003. PMID 12944502
- [Background] Jiang Y, Jahagirdar BN, Reinhardt RL, Schwartz RE, Keene CD, Ortiz-Gonzalez XR, Reyes M, Lenvik T, Lund T, Blackstad M, Du J, Aldrich S, Lisberg A, Low WC, Largaespada DA, Verfaillie CM. Pluripotency of mesenchymal stem cells derived from adult marrow. Nature. 2002 Jul 4;418(6893):41-9. doi: 10.1038/nature00870. Epub 2002 Jun 20. PMID 12077603
- [Derived] Davatchi F, Nikbin B, Shams H, Sadeghi Abdollahi B, Mohyeddin M, Shahram F. Mesenchymal stem cell therapy unable to rescue the vision from advanced Behcet's disease retinal vasculitis: report of three patients. Int J Rheum Dis. 2013 Apr;16(2):139-47. doi: 10.1111/1756-185X.12068. PMID 23773637